CLINICAL TRIAL: NCT01957670
Title: Pilot, Open-label, Single-Arm Study Designed to Clinically Evaluate Various Lacrima Medical Device Prototypes in Adult Patients With Dry Eye Syndrome
Brief Title: Pilot Study to Clinical Evaluate Device Prototypes in Dry Eye Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision due to change the clinical indication to Chronic Insomnia
Sponsor: Lacrima Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM001
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Dry Eye Syndrome
Keywords: Keratoconjunctivitis Sicca; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Lacrima medical device (Experimental)
  Interventions: Device: Lacrima medical Prototypes

INTERVENTIONS:
Device: Lacrima medical Prototypes

SUMMARY:
The study will assess the safety, tolerability and feasibility of Lacrima investigational medical device to treat dry eye patients

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female, 18 years of age and over at screening
2. Diagnosis of mild to moderate Dry Eye, as defined by:

   1. Positive corneal fluorescein staining , defined as a corneal punctate fluorescein staining score of ≥3 in either eye by the National Eye Institute evaluation scale summed over 5 areas, each with a 0-3 scoring scale; AND
   2. Schirmer Test score (with anesthesia, 5 minutes < 5 mm either eye) ; AND
   3. OSDI score of ≥12 and OSDI score of <33

Main Exclusion Criteria:

1. Persistent intraocular inflammation or infection including conjunctivitis at the time of the study or 2 weeks prior to study start.
2. Any concomitant active or history of eye disease including, but not limited to lid abnormalities, nasolacrimal obstruction, active ulcer, glaucoma or ocular herpes simplex virus infection
3. Patients currently using topical steroidal or anti-inflammatory eye drops for 1 month prior to screening
4. Receipt of any type of topical artificial eye drops within 3 days prior to screening
5. Receipt of topical cyclosporine eye drops within 3 months prior to screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Lower Tear Meniscus Height using Optical Coherence Tomography | up to 8 hours

SECONDARY OUTCOMES:
Visual Analog Scale score | up to 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Israel, Tel Aviv, Israel